CLINICAL TRIAL: NCT01027832
Title: Antibiotic Treatment in Ventilator Associated Tracheobronchitis (VAT): A Randomized, Controlled Trial
Brief Title: Antibiotic Treatment in Ventilator Associated Tracheobronchitis (VAT)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Arie Soroksky M.D., AGeneral ICU, Assaf Harofe MC, Zerifin 70300, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102/09
Record Dates: First submitted 2009-11-26; First posted 2009-12-09 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Tracheobronchitis
Keywords: tracheobronchitis
MeSH Terms: interventions — Piperacillin; Tazobactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm (No Intervention): no intervention
- Experimental arm (Experimental): antibiotics
  Interventions: Drug: Piperacillin/Tazobactam for 7 days

INTERVENTIONS:
Drug: Piperacillin/Tazobactam for 7 days — Piperacillin/Tazobactam for 7 days
  Arms: Experimental arm

SUMMARY:
Mechanically Ventilated patients in the intensive care unit (ICU) often present with fever, and purulent sputum, but without radiological evidence of pneumonia.

These patients may have tracheobronchitis. Some suspect that this condition precedes the development of pneumonia. Antibiotic treatment in tracheobronchitis is controversial.

The investigators will recruit patients with tracheobronchitis and randomize them into 2 groups. One group will be treated with antibiotics and the other group will serve as control.

DETAILED DESCRIPTION:
Patients with proved tracheobronchitis who are mechanically ventilated for more than 48 hrs, will undergo a CT scan to rool our pneumonia that may not be seen on a routine chest x-ray.

After ruling out pneumonia by CT scan, patients will be randomized into 2 groups. Intervention group will receive 7 days of treatment with Piperacillin/Tazobactam. A control group will receive nothing.

Primary endpoint wil be the rate of new pneumonias and secondary endpoint will be ICU Length of stay, days on mechanical ventilation and 28 day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Tracheobronchitis as defined by:

  * Purulent sputum with > 10 x 4 CFU
  * Leukocytosis or leukopenia
  * Fever
  * No pneumonia on CT scan

Exclusion Criteria:

* Recent treatment of pneumonia
* Abnormal Chest X-ray
* Evidence of Pneumonia on CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Rate of development of new pneumonia | 2 years

SECONDARY OUTCOMES:
ICU length of stay (LOS) and mortality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Arie Soroksky, MD, Principal Investigator — Tel Aviv University, Faculty of Medicine, Israel.
Locations (1):
- Assaf Harofe MC, Beer Yakov, Zerifin, Israel